CLINICAL TRIAL: NCT07373158
Title: Acute Modulation of Post-Exercise Recovery Through Inspiratory Muscle Activation in Professional Male Football Players: A Randomized Clinical Trial
Brief Title: Inspiratory Muscle Activation and Post-Exercise Recovery in Professional Football Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 021
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sports Physical Therapy; Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phrenic Electrostimulation (Experimental): The participant will be placed in the supine position, and the intervention will be performed using a pen-type electrode. Bilateral stimulation of the phrenic nerves will be applied below the sternal portion of the sternocleidomastoid muscle at the C3-C5 level. The electrical stimulators will be set to a mean frequency of 50 Hz and a pulse width of 300 μs. Stimulation intensity will be progressively increased until a visible diaphragmatic contraction (abdominal movement) is observed and reaches the maximum level tolerable for the player.
  The stimulation protocol will consist of two sets of 30 repetitions, delivered in bilateral cycles of 6 s ON (stimulation) and 10 s OFF (rest), including a 2-minute rest period between sets. Concurrently with the perception of the involuntary contraction, the participant will perform a voluntary contraction through diaphragmatic inspiration.
  Interventions: Device: Inspiratory muscle activation via phrenic nerve modulation
- Inspiratory muscle warm-up group (Active Comparator): Participants will breathe against submaximal inspiratory loads following a protocol consisting of two sets of 30 breaths, equivalent to 40% of their MIP, using the Breathcare MIP/MEP device (Big Breathe®, GH Innotek Co., Ltd., Busan, Republic of Korea). Breathing will be performed using a self-paced pattern, provided that a ratio of approximately 1 s of inspiration to 2 s of expiration is maintained to avoid hyperventilation.
  The session duration will correspond to the exact time required to complete the two sets of breaths, including a 2-minute rest period between sets, with an estimated total duration of approximately 15 minutes.
  Interventions: Device: Inspiratory muscle activation via threshold device
- Control group (No Intervention): Participants in this group will remain seated at rest in a quiet and controlled environment. During this period, they will breathe normally. The rest duration for this group will be identical to that of the other interventions.

INTERVENTIONS:
Device: Inspiratory muscle activation via phrenic nerve modulation — Phrenic nerve stimulation using low-frequency symmetric biphasic current
  Arms: Phrenic Electrostimulation
Device: Inspiratory muscle activation via threshold device — Deep inspirations against submaximal inspiratory load
  Arms: Inspiratory muscle warm-up group

SUMMARY:
Respiratory muscles play a fundamental role in sports performance. Fatigue of these muscles induces changes in maximal inspiratory pressure and autonomic nervous system activity, thereby compromising the athlete's recovery process. The primary aim of this study is to evaluate the specific effects of different inspiratory muscle activation modalities on post-exercise recovery in professional male football players. The study seeks to determine which of the three modalities-bilateral phrenic nerve electrical stimulation, a threshold loading device protocol, or inactivity-provides greater benefits for recovery. The effectiveness of these interventions will be assessed using two key outcome variables: maximal inspiratory pressure (MIP) and heart rate variability (HRV).

This study is designed as a randomized clinical trial (RCT) in which participants will be allocated into three intervention groups: a bilateral phrenic nerve electrical stimulation group (EG1), in which involuntary diaphragmatic contractions will be induced using an electrotherapy device with current applied to the phrenic nerves; a threshold device group (EG2), in which participants will perform breathing against submaximal inspiratory loads equivalent to 40% of their MIP; and a control group (CG), which will remain seated for a period equivalent to the duration of the other interventions. Group allocation will be ensured through randomization using Microsoft Excel.

Regarding statistical analysis, data normality will be assessed using the Shapiro-Wilk test. Comparisons of quantitative variables will be performed using Student's t test when normality assumptions are met, or the Mann-Whitney U test otherwise. A p value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Male professional football player.
* Currently under an active professional contract and participating in regular competition.
* Aged between 18 and 40 years.
* No participation in inspiratory muscle training (IMT) programs in the past 12 months.
* Signed informed consent provided by the participant.

Exclusion Criteria:

* Musculoskeletal injuries or surgical interventions within the past 6 months.
* Use of medications affecting cardiac or respiratory function (e.g., beta-blockers, beta-adrenergic inhibitors).
* Presence of any acute and/or chronic disease (cardiorespiratory, neurological, metabolic, oncological, etc.).
* Use of tobacco, recreational drugs, or stimulant substances.
* Metallic implants in the cervical region.
* Presence of a pacemaker.
* Current participation in other inspiratory muscle training programs.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Hear rate variability | Pre-match 24 hours before (baseline); Post-match 24 hours (pre-intervention); Immediately post-intervention; 15 minutes post-intervention; 30 minutes post-intervention
  HRV will be assessed using a heart rate monitor (Polar H10; Polar Electro Oy, Kempele, Finland) with participants in the supine position in a quiet room (~25 °C, dim lighting). Cardiac signals will be recorded for 3 minutes via a chest strap. Participants will avoid caffeine, alcohol, tobacco, and intense exercise for 12 h prior, and refrain from speaking or voluntary movements during recording. Analysis will be performed with Kubios HRV 3.1.0 (University of Kuopio, Finland), examining LF/HF ratio, LF (0.04-0.15 Hz) and HF (0.15-0.40 Hz) power in normalized units, SDNN, and RMSSD.

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure | Pre-match 24 hours before (baseline); Post-match 24 hours (pre-intervention); Immediately post-intervention; 15 minutes post-intervention; 30 minutes post-intervention
  Maximal inspiratory pressure (MIP) will be assessed with participants in a seated position using the Breathcare MIP/MEP device (Big Breathe®, GH Innotek Co., Ltd., Busan, Republic of Korea). The examiner will demonstrate the maneuver prior to its execution. To ensure proper airflow through the mouth, the nostrils will be occluded. Participants will perform up to six maneuvers per attempt, with a 1-minute rest between each. The most consistent and reproducible result from three attempts, with a variation of less than 5%, will be selected for analysis.

IPD SHARING:
Plan to Share IPD: Yes
The availability of the data, and the materials will be available at the request of the publisher.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code